CLINICAL TRIAL: NCT00130312
Title: The Collaborative Study Group Trial: The Effect of Sulodexide in Overt Type 2 Diabetic Nephropathy
Brief Title: Effect of Sulodexide in Overt Diabetic Nephropathy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No difference in protein excretion at 6&12 months. No safety issues.
Sponsor: Keryx Biopharmaceuticals (Industry)
Collaborators: Collaborative Study Group (CSG) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KRX-101-401; NCT00342238 (obsolete NCT alias)
Record Dates: First submitted 2005-08-11; First posted 2005-08-15 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetes; Diabetic Nephropathy; Proteinuria
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Proteinuria | interventions — glucuronyl glucosamine glycan sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sulodexide (Experimental): Also known as KRX-101. These patients are also on ACEs and ARBs (irbesartin and/or losartan).
  Interventions: Drug: Sulodexide
- Placebo (Placebo Comparator): These patients are also on ACEs and ARBs (irbesartin and/or losartan).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sulodexide — 100 mg gelcap in the morning and evening
  Other Names: KRX-101
  Arms: Sulodexide
Drug: Placebo — 1 placebo gelcap in the morning and evening
  Other Names: placebo gelpcap
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether sulodexide is effective in slowing or preventing the progression of diabetic kidney disease.

DETAILED DESCRIPTION:
Diabetes is now the most common cause of end-stage renal disease (ESRD) in the U.S. and in many other developed nations. Diabetic nephropathy now represents 44% of all new cases of ESRD in the U.S. Despite advances in clinical care, including improvements in glycemic and blood pressure control, the number of new cases of diabetes related ESRD continues to rise. In particular, the incidence of type 2 diabetes mellitus (DM2)-related cases of ESRD is rapidly increasing. From 1993 to 1997, 71% of all diabetes-related ESRD was attributable to DM2 (USRDS 1999). The earliest sign of diabetic kidney disease presents as microalbuminuria, the spilling of small of amounts of blood protein into the urine. Microalbuminuria correlates directly with the subsequent development of more advanced kidney disease. Improved glycemic control and blood pressure control with the use of inhibitors of the renin-angiotensin-aldosterone system can reduce the level of microalbuminuria and overt proteinuria. However, despite these measures, diabetic nephropathy continues to progress, albeit more slowly. Sulodexide belongs to a class of drugs called glycosaminoglycans (GAG). GAG therapy has been shown in animal models to prevent and or induce regression of albuminuria, and the morphologic changes associated with progressive diabetic nephropathy such as glomerular basement thickening, loss of the anionic charge density and mesangial collagen deposition. Sulodexide is approved in Europe to treat vascular indications. It has been utilized in several small phase II studies to treat early diabetic nephropathy, inducing an additional 40-70 % reduction in albuminuria in subjects whose albumin excretion was already reduced with tight glycemic control plus the use of inhibitors of the renin-angiotensin-aldosterone system for blood pressure control.

The purpose of this study is to add to this body of evidence that Sulodexide may offer additional benefit in preventing or ameliorating more advanced diabetic nephropathy manifested as overt proteinuria and reduced GFR. Subjects with type 2 diabetes, moderately elevated serum creatinine and overt proteinuria will be treated with a standardized maximal recommended/tolerated dose of irbesartan 300 mg/day or losartan 100 mg/day plus additional concomitant non-ARB, non-ACEi antihypertensive drugs,for up to 2-3 months to establish adequate and stable blood pressure control and urine protein excretion. After establishing baseline serum creatinine and urine protein excretion they will be randomized to either Sulodexide 200 mg/d or matching placebo. Subjects will be seen every 3 months to monitor safety and efficacy parameters for up to 4 years. The primary outcome is a doubling of baseline serum creatinine (50% loss of kidney function) or end stage kidney disease (ESRD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes;
* Urine protein to creatinine ratio (PCR) equal to or greater than 900 mg/G (101.7 mg/mmol) in women and equal to or greater than 650 mg/G (73.45 mg/mmol) in men;
* Serum creatinine in women 1.3 - 3.0 mg/dL (115-265 μmol/L), inclusive, and in men 1.5 - 3.0 mg/dL (133-265 μmol/L), inclusive;
* Willing to discontinue antihypertensive medication regimen, if applicable;
* Willing and able to give informed consent.

Exclusion Criteria:

* Type 1 (insulin-dependent; juvenile onset) diabetes;
* Renal disease as follows:

  * Patients with known non-diabetic renal disease (nephrosclerosis superimposed on diabetic nephropathy acceptable), or
  * Renal allograft;
* Absolute requirement for combination therapy of angiotensin converting enzyme inhibitors (ACEI) and angiotensin receptor blockers (ARB);
* Patients who require ACEI, but not ACEI/ARB combination;
* Cardiovascular disease as follows:

  * Unstable angina pectoris within 3 months of study entry;
  * Myocardial infarction, coronary artery bypass graft surgery, or percutaneous transluminal coronary angioplasty/stent within 3 months of study entry;
  * Transient ischemic attack within 3 months of study entry;
  * Cerebrovascular accident within 3 months of study entry;
  * New York Heart Association Functional Class III or IV (Note: if a patient is New York Heart Association Functional Class I or II and requires an ACEI, consult with the Clinical Coordinating Center to obtain permission for the patient to be on an ACEI rather than an ARB);
  * Obstructive valvular heart disease or hypertrophic cardiomyopathy; or
  * Second or third degree atrioventricular block not successfully treated with a pacemaker;
* Need for chronic (>2 weeks) immunosuppressive therapy, including corticosteroids (excluding inhaled or nasal steroids);
* New diagnosis of cancer or recurrent cancer within 5 years of screening (except non-melanoma skin cancer);
* Psychiatric disorder that interferes with the patient's ability to comply with the protocol;
* Inability to tolerate oral medication or a history of significant malabsorption;
* History of alcohol or other drug abuse within 12 months of study entry;
* Known human immunodeficiency virus disease;
* Any other medical condition which renders the patient unable to or unlikely to complete the study, or which would interfere with optimal participation in the study or produce significant risk to the patient;
* Receipt of any investigational drugs (including placebo) within 30 days of enrollment;
* Evidence of hepatic dysfunction including total bilirubin >2.0 mg/dL (>35 micromol/L) or liver transaminase (aspartate aminotransferase [AST] or alanine transferase [ALT]) >3 times upper limit of normal;
* Anticipate need for surgery;
* Inability to cooperate with study personnel or history of noncompliance to medical regimen;
* Known allergies or intolerance to any heparin-like compound including heparin-induced thrombocytopenia Type II;
* Prior exposure to sulodexide, either in a clinical setting or as a participant in another clinical study.
* Untreated urinary tract infection that would impact urinary protein values.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 968 (Actual)
Dates: Start 2005-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Time to doubling of the serum creatinine or end stage kidney disease (ESRD) | Time in study depended on time to doubling of serum creatinine
  Time in study depended on time to doubling of serum creatinine and when the patient was enrolled in the trial.
Safety and tolerance of sulodexide therapy long-term | Time in study depended on time to doubling of serum creatinine
  Review of laboratory parameters, adverse events, physical examinations, etc. were made to evaluate patient safety.

SECONDARY OUTCOMES:
Change in urinary protein/albumin excretion | Time in study depended on time to doubling of serum creatinine
  Review of urinary protein and albumin excretion was made as an additional assessment of kidney function.

CONTACTS AND LOCATIONS:
Overall Officials: Edmund J Lewis, MD, Study Director — The Collaborative Study Group, Rush University Medical Center, Chicago, IL USA; Robert C Atkins, M.D., Principal Investigator — The Collaborative Study Group, Monash Medical Center, Clayton, Victoria, AUSTRALIA; Dick deZeeuw, M.D., Principal Investigator — The Collaborative Study Group, University of Groningen, NETHERLANDS; Itamar Raz, M.D., Principal Investigator — The Collaborative Study Group, Hadassah University, Jerusalem, ISRAEL
Locations (3):
- The Collaborative Study Group, Clinical Coordinating Center for U.S. and Canadian clinics, Rush University Medical Center, Chicago, Illinois, United States
- The Collaborative Study Group, Clinical Coordinating Center for the Pacific Region, Monash Medical Center, Melbourne, Victoria, Australia
- The Collaborative Study Group, Clinical Coordinating Center for European Clinics, University of Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bidadkosh A, Lambooy SPH, Heerspink HJ, Pena MJ, Henning RH, Buikema H, Deelman LE. Predictive Properties of Biomarkers GDF-15, NTproBNP, and hs-TnT for Morbidity and Mortality in Patients With Type 2 Diabetes With Nephropathy. Diabetes Care. 2017 Jun;40(6):784-792. doi: 10.2337/dc16-2175. Epub 2017 Mar 24. PMID 28341782